CLINICAL TRIAL: NCT01798316
Title: IV Acetaminophen for Postoperative Analgesia After Laparoscopic Cholecystectomy
Brief Title: IV Acetaminophen for Postoperative Analgesia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Principal Investigator left the institution
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-0409; IRB #12-409B (Other: North Shore-Long Island Jewish Health System)
Record Dates: First submitted 2013-02-05; First posted 2013-02-25 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Postoperative Pain; Postoperative Nausea; Postoperative Vomiting
Keywords: IV Acetaminophen; Laparoscopic cholecystectomy; Postoperative nausea; Postoperative vomiting
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Acetaminophen; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Acetaminophen (Active Comparator): IV Acetaminophen administered on admission to post-anesthesia care unit
  Interventions: Drug: IV Acetaminophen
- Standard of care (Active Comparator): Standard of care pain management regimen including opioids administered on admission to post-anesthesia care unit
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: IV Acetaminophen — Single dose, 1000g mg infusion over 15 minutes plus standard of care pain management regimen
  Other Names: Ofirmev
  Arms: IV Acetaminophen
Drug: Standard of Care — Standard of care pain management regimen, no IV Acetaminophen,
  Other Names: As per provider: Opioids
  Arms: Standard of care

SUMMARY:
The purpose of this study is to evaluate the use of IV acetaminophen for postoperative pain management after laparoscopic cholecystectomy to determine if its use to supplement standard of care pain management decreases the incidence of post-operative nausea and vomiting.

DETAILED DESCRIPTION:
The recent clinical development of an intravenous (IV) acetaminophen formulation for use in the US has important implications for the management of postoperative pain given its safety profile and suitability for use in the early phase of the postoperative period. In clinical studies a significant opioid-sparing effect has been documented with a substantial percentage of patients avoiding the need for opioid rescue medication altogether. This avoidance or delay in the use of opioids has been shown to reduce undesirable side effects. It is proposed that the use of IV acetaminophen in the post anesthesia care unit (PACU) for postoperative analgesia after laparoscopic cholecystectomy will result in decreased incidence of post operative nausea and vomiting (PONV) and decreased use of narcotics.

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing pre-scheduled laparoscopic cholecystectomy;
* American Society of Anesthesiology patient classification status I-II

Exclusion Criteria:

* Regular preoperative use of or opioids,
* Subjects admitted after surgery for postoperative complications other than postoperative pain or PONV.
* Subjects converted to open laparoscopic cholecystectomy
* Known allergy/hypersensitivity to acetaminophen
* Use of opioids prior to commencement of the study (<7 days)
* Patients with chronic pain conditions or disease requiring pain control
* Abnormal liver function
* Known or suspected alcohol, drug or opiate abuse or dependence
* Patients with a BMI of greater than 35
* Other physical, mental or medical conditions that could effect participation.
* Abnormal renal function; serum creatinine>2gm/dl

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank J Overdyk, MD, Principal Investigator — Northwell Health
Locations (3):
- United States (3):
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Syosset Hospital, Syosset, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Acetaminophen: IV Acetaminophen administered before PACU admission
  IV Acetaminophen: Single dose, 1000g mg infusion over 15 minutes
- Standard of Care: Standard of care pain management regimen including opioids
  Standard of Care: without IV acetaminophen
Period: Overall Study
Arm/Group | IV Acetaminophen | Standard of Care
Started | 52 | 53
Completed | 52 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care: Standard of care pain management regimen including opioids
  Standard of Care: No IV acetaminophen
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen | Standard of Care | Total
Number analyzed (Participants) | 52 | 53 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (13.0) | 44.9 (12.3) | 44.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 12 | 13 | 25
Region of Enrollment [Number; unit: participants]
  United States | 52 | 53 | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Nausea and Vomiting (PONV).
Description: Number of participants with postoperative nausea and vomiting (PONV) will be recorded during PACU stay.
  PONV is defined as nausea intensity of 4 or higher on 0-10 numeric rating scale (NRS) and/or at least one episode of vomiting/retching.
Time Frame: 4 hours plus/minus 30 minutes
Measure: Count of Participants; unit: Participants
Groups:
- IV Acetaminophen: IV Acetaminophen administered on admission to PACU
  IV Acetaminophen: Single dose, 1000g mg infusion over 15 minutes plus standard of care
- Standard of Care: Standard of care pain management regimen including opioids administered on admission to PACU
  No IV Acetaminophen
Arm/Group | IV Acetaminophen | Standard of Care
Number analyzed (Participants) | 52 | 53
Participants | 15 | 17
Statistical Analysis 1: Comparison: IV Acetaminophen vs Standard of Care; Test type: Superiority or Other; p > 0.05, Chi-squared

2. Secondary Outcome: Number of Participants With Post Discharge Nausea and Vomiting (PDNV)
Description: Number of participants reporting post discharge nausea and vomiting (PDNV) documented up to 2 days following surgery.
  PDNV is defined as nausea intensity of 4 or higher on 0-10 numeric rating scale (NRS) and/or at least one episode of vomiting/retching following discharge.
Time Frame: Up to two days following surgery
Population: Post-discharge follow up group. Patients not included in analysis were lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | Standard of Care
Number analyzed (Participants) | 41 | 40
Participants | 4 | 10

3. Secondary Outcome: Highest Pain Intensity Score Using Numeric Rating Scale (NRS)
Description: Highest pain intensity reported during PACU stay using a 11-point (0-10) pain intensity numeric rating scale (NRS). Higher values represent higher pain intensities.
Time Frame: 4 hours plus/minus 30 minutes
Measure: Median (Inter-Quartile Range); unit: Units on a numerical rating scale
Groups:
- IV Acetaminophen: IV Acetaminophen administered before PACU admission
  IV Acetaminophen: Single dose, 1000g mg infusion over 15 minutes plus standard of care
Arm/Group | IV Acetaminophen | Standard of Care
Number analyzed (Participants) | 52 | 53
Units on a numerical rating scale | 6 [5 to 8] | 6 [4 to 8]

4. Secondary Outcome: Patient Satisfaction on a 5 Point Likert Scale
Description: Number of patients very satisfied or satisfied with pain and PONV management during hospital stay
Time Frame: Up to one week following surgery
Population: Post-discharge follow up group. Patients not included in analysis were lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | Standard of Care
Number analyzed (Participants) | 41 | 40
Participants | 38 | 35

5. Secondary Outcome: Pain Intensity Score 1 Hour Following Surgery Using Numeric Rating Scale
Description: Pain intensity score reported by participants 1 hour following surgery using an 11-point, 0-10 Numeric Rating Scale (NRS). Higher scores indicate higher pain intensities
Time Frame: 1 hour following surgery
Measure: Median (Inter-Quartile Range); unit: Units on a numerical rating scale
Arm/Group | IV Acetaminophen | Standard of Care
Number analyzed (Participants) | 52 | 53
Units on a numerical rating scale | 3 [0 to 4] | 3 [0 to 4]

6. Other Pre Specified Outcome: Number of Patients Requiring Rescue Analgesia for Breakthrough Pain
Description: Number of patients requiring rescue analgesia medication during first hour of PACU stay
Time Frame: 1 hour following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | Standard of Care
Number analyzed (Participants) | 52 | 53
Participants | 28 | 20

7. Other Pre Specified Outcome: Narcotic Use During PACU Stay
Description: Narcotic medication administered during PACU stay in morphine milligram equivalents
Time Frame: 4 hours plus/minus 30 minutes
Measure: Mean (95% Confidence Interval); unit: Morphine milligram equivalents
Arm/Group | IV Acetaminophen | Standard of Care
Number analyzed (Participants) | 52 | 53
Morphine milligram equivalents | 13.3 [8.5 to 18.0] | 16.8 [10.3 to 23.2]

ADVERSE EVENTS:
Arm/Group | IV Acetaminophen | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/53
Other Adverse Events (participants affected / at risk) | 18/52 | 23/53
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IV Acetaminophen (N=52) | Standard of Care (N=53)
Nausea (Gastrointestinal disorders) | 10 | 15
Drowziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes